#### Appendix A Protocol

#### **Investigator-Initiated Study Protocol**

In Clinic Optometrist Insertion of Dextenza Prior to Cataract Surgery

### The PREPARE Study

Compound: DEXTENZA (dexamethasone

ophthalmic insert) 0.4 mg, for

intracanalicular use

Study Name: In Clinic Optometrist Insertion of

Dextenza Prior to Cataract Surgery

The Prepare Study

Clinical Phase: Investigator-Initiated Clinical Trial

**Date of Issue:** 9/24/2020

Primary Investigator: Mitch Ibach, OD

Sub Investigator: Justin Schweitzer, OD

John Berdahl, MD Doug Wallin, OD Keith Rasmussen, OD Vance Thompson, MD Larae Zimprich, OD Jason Schmit, OD Daniel Terveen, MD

Site Name & Location: Vance Thompson Vision Center

3101 West 57<sup>th</sup> Street Sioux Falls, South Dakota

57108

| CLINICAL STUDY PROTO | |
|---|---|
| TITLE | The PREPARE Study |
| SITE LOCATION(S) | Vance Thompson Vision Center |
| | 3101 West 57th Street |
| | Sioux Falls, South Dakota |
| Daniegra | 57108 |
| PRINCIPAL | Mitch Ibach, OD |
| INVESTIGATOR | m 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| OBJECTIVE(S) | To evaluate the clinical outcomes with optometrist |
| | pre-surgical insertion of DEXTENZA in the clinical |
| | office setting in patients undergoing same-day |
| | cataract surgery compared to standard of care |
| | steroid therapy. |
| STUDY DESIGN | Prospective Open-label Interventional Study |
| STUDY DURATION | 2-3 months from start-up |
| ESTIMATED STUDY | Insert date of study completion |
| COMPLETION DATE | |
| POPULATION | |
| Sample Size: | N=60 (30 patients, 60 eyes) |
| Target Population: | Patients planning to undergo sequential bilateral |
| | cataract surgery. |
| TREATMENT(S) | |
| Study Drug | DEXTENZA (dexamethasone ophthalmic insert) 0.4 |
| • • | mg, for intracanalicular use |
| Dose/Route/Schedule: | All patients will be enrolled for cataract surgery. |
| | Each study subject will have their first eye |
| | randomized to either the Control Group or the |
| | Experimental Group. The second eye will be selected |
| | for the opposite group. All eyes will receive |
| | intracameral |
| | dexamethasone+moxifloxacin+ketorolac (DMK) at |
| | the time of surgery. All eyes will be placed on topical |
| | antibiotic (Vigamox 0.5%) QID for one week and |
| | topical NSAID ((Prolensa (Bromfenac 0.07%)) QD for |
| | one month. |
| | T |
| | Experimental Group (Treatment A): 30 eyes will |
| | receive DEXTENZA insertion, placed in the office by |
| | the optometrist prior to their same-day cataract |
| | surgery. |
| | Control Group (Treatment B): 30 eyes will receive |
| | Convict Group (Troublette D). 50 Cycs will receive |

topical prednisolone acetate 1% QID for one week, TID for one week, BID for one week, QD for one week.

## ENDPOINT(S) Primary:

To determine the effect of dexamethasone intracanalicular insert through Week 4 as measured bv:

- Mean anterior chamber cell/flare score as measured by Slit Lamp Biomicroscopy evaluation using grading scale of 0 to 4 + (SUN Working Group Grading Scheme) at post-op Day 1, Day 7, and Week 4.
- Mean pain score as measured by Visual Analog Score numerical grading scale 0-10 at post-op Day 1, Day 7, and Week 4.

To determine patient preference through Week 4 as measured by:

- Adapted COMTOL Questionnaire at Week 4. To determine the effect of dexamethasone intracanalicular insert through Week 4 or 12:
  - Incidence of increased intraocular pressure (IOP) >10mmHg above baseline as measured by Goldmann Applanation Tonometer at postop Day 1, Day 7, and Week 4.
  - Incidence of Cystoid Macular Edema (CME) as measured by optical coherence tomography (OCT) at post-op Week 4.

To determine physician ease of insertion following dexamethasone intracanalicular insert placement prior to same-day surgery as measured by:

Physician Ease of Use Survey following dexamethasone intracanalicular placement on Surgical Visit Day 0.

To determine eye drop therapy burden on the patient through Week 4 as measured by:

Eye Drop Burden Questionnaire at post-op Day 7 and Week 4.

#### Secondary:

#### TABLE OF CONTENTS

| | linical Study Protocol Synopsisist of Tables | |
|----|----------------------------------------------------|----|
| | Introduction and Rationale | |
| Ι. | 1.1 Introduction | |
| | 1.2 Rationale | |
| | 1.2.1 Rationale for Study Design | |
| 2 | Study Objectives | |
| | 2.1 Primary Objective | |
| | 2.2 Secondary Objectives | |
| 3. | Study Design | |
| | 3.1 Study Description and Duration | |
| 4. | Selection, Withdrawal, and Replacement of Patients | |
| | 4.1 Study Population | |
| | 4.1.1 Inclusion Criteria | 26 |
| | 4.1.2 Exclusion Criteria | 26 |
| | 4.2 Treatment Logistics and Accountability | 27 |
| | 4.2.1 Packaging, Labeling, and Storage | |
| | 4.2.2 Supply and Disposition of Treatments | |
| | 4.2.3 Treatment Accountability | |
| | 4.3 Concomitant Medications and Procedures | |
| 5. | Study Schedule of Events and Visit Descriptions | |
| | 5.1 Schedule of Events | |
| | 5.2 Study Visit Descriptions | |
| | 5.2.1 Study Procedures | |
| | 5.2.2 Unscheduled Visits | |
| | 5.2.3 Adverse Event Information Collection | |
| c | 5.3 Rescue Criteria | |
| 6. | v / 1 0/ 0 | |
| | 6.1 Definitions | |
| | 6.1.1 Adverse Event | |
| | 6.2 Recording and Reporting Adverse Events | |
| 7 | Study Variables | |
| ١. | 7.1 Demographic and Baseline Characteristics | |
| 8 | Ethical and Regulatory Considerations | |
| Ο. | 8.1 Good Clinical Practice Statement | |
| | 8.2 Informed Consent | |
| | 8.3 Patient Confidentiality and Data Protection | |
| | 8.4 Institutional Review Board | |
| | | - |
| | T | |

#### LIST OF TABLES

Table 1 Schedule of Events ...... 

#### Introduction and Rationale

#### Introduction

Dextenza (dexamethasone 0.4mg ophthalmic insert) is a steroid eluting intracanalicular plug approved on-label for the treatment of pain and postoperative inflammation in patients who've undergone ocular surgery. Utilizing Dextenza, in place of ophthalmic steroid drops, will provide patients with a lessened number of postoperative drops which decreases both contamination possibilities and improper drug installation. Dextenza's hydrogel technology is proposed to offer patients a gradual sustained delivery of steroid to the ocular surface which may decrease subjective postoperative pain.

Post-operative drop regimens frequently induce both concerns and questions for patients undergoing ocular surgery. Poor compliance with postoperative medications can lead to unexpected and or unsatisfactory outcomes. In post-operative cataract surgery patients, un-treated or non-resolving inflammation can lead to pain, anterior chamber inflammation, and potentially cystoid macular edema (CME). Lessening the risk of these adverse events due to drop complications is a key benefit of Dextenza. There may be future possibilities to combine intracameral medication combinations (antibiotic, steroid, NSAID) plus Dextenza to further reduce the patient post-operative drop burden.

On introduction to the market, Dextenza was most commonly inserted in the operating room (OR) pre-cataract surgery, but other instillation protocols will increase practitioner adoption and patient access. Increasing optometrist administration in clinic allows for another route for insurance reimbursement while freeing up ophthalmologists in the OR.

#### Rationale

DEXTENZA (dexamethasone 0.4mg ophthalmic insert) has increasing research and evidence for post-cataract surgery patients, but a gap remains in best practices for instillation timing and protocols. In clinic insertion provides another route for device administration which can help foster additional reimbursement codes.

Dextenza's ability to treat post-operative inflammation while also increasing remaining tear volume by punctal occlusion has potential to improve visual outcomes for patients while also decreasing post-operative drop inconvenience. The studied patient population is having their initial cataract evaluation and surgery on the same day, decreasing patient inconvenience, adding Dextenza is another arrow in the quiver.

## Rationale for Study Design

This prospective contralateral eye study will compare the outcomes of 30 patients undergoing cataract surgery. All eyes will receive intracameral DMK at the conclusion of surgery. All eyes will be treated with Vigamox 0.5% QID for 1 week and Prolensa

(bromfenac 0.07%) QD for 1 month. After randomization, one eye per patient will receive Dextenza in place of topical steroid while the other eye has topical prednisolone acetate 1% QID 1 week, TID 1 week, BID 1 week, and QD 1 week. The primary endpoints of anterior chamber cell and mean pain score correlate to the initial FDA approval trial for Dextenza. The study inclusion and exclusion criteria were chosen based on patients who normally would be successful with cataract surgery, including the absence of pre-existing intraocular inflammation or macular edema. The study follow-up visits were based on the Vance Thompson Vision standard postoperative follow-up protocols.

#### Study Objectives

## **Primary Objective**

To determine the effect of dexamethasone intracanalicular insert through Week 4 as measured by:

- Mean anterior chamber cell score as measured by Slit Lamp Biomicroscopy evaluation using grading scale of 0 to 4 + (SUN Working Group Grading Scheme) at post-op Day 1, Day 7, and Week 4.
- Mean pain score as measured by Visual Analog Score numerical grading scale 0-10 at post-op Day 1, Day 7, and Week 4.

To determine patient preference through Week 4 as measured by:

• Adapted COMTOL Questionnaire at Week 4.

## Secondary Objectives

To determine the effect of dexamethasone intracanalicular insert through Week 4 or 12:

- Mean anterior chamber flare score as measured by Slit Lamp Biomicroscopy evaluation using grading scale of 0 to 4 + (SUN Working Group Grading Scheme) at post-op Day 1, Day 7, and Week 4.
- Incidence of increased intraocular pressure (IOP) >10mmHg above baseline as measured by Goldmann Applanation Tonometer at post-op Day 1, Day 7, and Week 4.
- Incidence of Cystoid Macular Edema (CME) as measured by optical coherence tomography (OCT) at post-op Week 4.

To determine physician ease of insertion following dexamethasone intracanalicular insert placement prior to same-day surgery as measured by:

• Physician Ease of Use Survey following dexamethasone intracanalicular placement on Surgical Visit Day 0.

To determine eye drop therapy burden on the patient through Week 4 as measured by:

• Eye Drop Burden Questionnaire at post-op Day 7 and Week 4.

## Study Design

## Study Description and Duration

This prospective, open-label, randomized, investigator-sponsored clinical study seeks to investigate a new protocol for in-clinic Dextenza insertion by optometrists at the day of surgery. This three month study will study the clearance of intraocular pain and inflammation comparing topical steroids versus Dextenza.

## Selection, Withdrawal, and Replacement of Patients Study Population

The study aims to enroll 30 patients undergoing routine sequential bilateral cataract surgery.

#### **Inclusion Criteria**

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

- Patients 18 years of age or older, undergoing routine, uncomplicated, sequential bilateral cataract surgery.
- Willing and able to comply with clinic visits and study related procedures
- Willing and able to sign the informed consent form

#### **Exclusion Criteria**

A patient who meets any of the following criteria will be excluded from the study:

- Patients under the age of 18.
- Patients who are pregnant (must be ruled out in women of child-bearing age with pregnancy test).
- Active infectious ocular or systemic disease.
- Patients with active infectious ocular or extraocular disease.
- Patients actively treated with local or systemic immunosuppression including systemic corticosteroids.
- Patients with known hypersensitivity to Dexamethasone.
- Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator.
- Patients with proliferative diabetic retinopathy or uncontrolled diabetes as deemed by an A1C > 10.0.
- Patients with a history of ocular inflammation or macular edema.
- Patients with a pre-existing epiretinal membrane (ERM)
- Patients with allergy or inability to receive intracameral antibiotic.
- Patients on systemic non-steroidal anti-inflammatory drugs (NSAID) greater than 1,200 mg/day

• Patients with a corticosteroid implant (i.e. Ozurdex).

# Treatment Logistics and Accountability Packaging, Labeling, and Storage

Intracanalicular dexamethasone insert must be stored in a secure area accessible only to the Investigator and their designee(s) and refrigerated and stored between 2° C and 8° C. Intracanalicular dexamethasone insert contains 0.4 mg dexamethasone and is designed to provide a sustained and tapered release of therapeutic levels of dexamethasone to the ocular surface for up to 30 days for the reduction of post-surgical inflammation and pain associated with ocular surgery. Dexamethasone is an anti-inflammatory 9-fluoro-glucocorticoid (also termed a glucocorticoid agonist) and is the active ingredient found in MAXIDEX® 0.1% (dexamethasone ophthalmic suspension), which contains approximately 50 µg of dexamethasone per drop.

Study inserts will be supplied by Ocular Therapeutix in a sealed foil pouch containing one intracanalicular dexamethasone insert in a foam carrier.

Study inserts will be shipped to the site via overnight shipping using cold packs to maintain a temperature of 2° to 8° C. The Investigator, or an approved representative (e.g. pharmacist), will ensure that all study drug inserts are stored in a secured area, under recommended storage conditions and in accordance with applicable regulatory requirements. The shipping box is to be opened and stored immediately at the site in a refrigerator intended for investigational products at a temperature of 2° to 8°C.

When the insert is removed from the refrigerator, it should be visually inspected. Exposure of the insert to temperatures outside these limits it not recommended. Records of actual storage conditions (i.e. temperature log) at the study site must be maintained; and must include a record of the dates, when the refrigerator was checked, the initials of person checking, and the temperature.

## Supply and Disposition of Treatments

Study insert will be shipped at a temperature of 2° to 8°C to the investigator as needed during the study.

## Treatment Accountability

All study insert accountability records will be kept current.

The investigator will account for all opened and unopened packaging of study inserts. These records will contain the dates, quantity, and study medication

- Inserted in each patient,
- disposed of at the site or returned to Ocular Therapeutix

All accountability records will be made available for inspection by regulatory agency inspectors.

## Concomitant Medications and Procedures

At the discretion of their physician, patients may continue to receive all medications and standard treatments administered for other conditions.

# Study Schedule of Events and Visit Descriptions Schedule of Events

Study assessments and procedures are presented by visit in Table 1 below.

Table 1 Schedule of Events

| Table 1 Schedule | of Event | /B | | 1 | 1 | | ı | | 1 |
|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Screening/<br>Baseline | First<br>Eye<br>Surgical<br>Visit<br>Day 0 | First<br>Eye<br>Day 1 | Second<br>Eye<br>Surgical<br>Visit<br>Day 0 | Second<br>Eye<br>Day 1 | Day 7<br>Both<br>Eyes | Day 30<br>Both<br>Eyes | Day 90<br>post-op<br>Both<br>Eyes | Early<br>Termination |
| Visit | VISIT 1 | VISIT 2 | VISIT 3 | VISIT 4 | VISIT 5 | VISIT | VISIT 7 | VISIT 8 | |
| Windows for Visits | (Day -30 to 0) | | | | | 6<br>+/- 2<br>day<br>from<br>first<br>eye sx | +/- 5<br>days<br>from<br>first eye<br>sx | +/- 7<br>days<br>from<br>first eye<br>sx | |
| Inclusion/Exclusion | X | | | | | | | | |
| Informed Consent | X | | | | | | | | |
| Demographics | X | | | | | | | | |
| Medical History and Concurrent Illnesses | X | X | X | X | X | X | X | X | |
| Concomitant Medications | X | X | X | X | X | X | X | X | |
| Uncorrected Distance VA | X | | X | | X | X | X | X | |
| MRX | X | | | | | X | X | X | |
| BCVA (ETDRS at 4m) | X | | | | | X | X | X | |
| Ophthalmic Examination (dilated fundus | X | | | | | | X | | |
| exam) Slit lamp exam | X | | X | | X | X | X | X | |
| Grade cataract density (scale 1 to 4) | | X | | X | | | | | |
| OCT | X | | | | | | X | | |
| Intraocular Pressure | X | | X | | X | X | X | X | |
| Indicate the incision type, location, and size (mm) | | X | | X | | | | | |
| Type of IOL (e.g. monofocal, toric, multifocal, etc.) and lens power | | X | | X | | | | | |
| Record any surgical complications | | X | | X | | | | | |
| Subject reported AEs prior to or after surgery | | X | X | X | X | X | X | X | |
| Intracanalicular dexamethasone insert<br>(*if randomized to Dextenza arm) | | X | | X | | | | | |
| Intracameral injection of<br>NSAID+antibiotic+steroid combo | | X | | X | | | | | |
| Physician Ease of Use Survey | | X | | X | | | | | |
| Eye Drop Burden Questionnaire | | | | | | X | X | | |
| Adapted COMTOL Questionnaire | | | | | | | X | | |
| Ocular Pain Assessment | X | | X | | X | X | X | X | |
| Anterior chamber cell count | X | | X | | X | X | X | X | |
| Anterior chamber cell flare | X | | X | | X | X | X | X | |
| Insert Visualization | | X | X | X | X | X | X | X | |
| Prescribe post-operative topical therapy<br>regimen (*specific to each study group) | | X | | X | | | | | |

## 5.2 Study Visit Descriptions

### 5.2.1 Study Procedures

#### Screening/Baseline

After the patient has provided informed consent, the following information will be collected (if the data was collected within 30 days of the screening exam it may be pulled forward from the subject previous exam):

- Inclusion/exclusion
- Demographics
- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- MRX
- BCVA
- Ophthalmic Examination (dilated fundus exam)
- Slit lamp Exam
- OCT
- IOP
- Ocular Pain Assessment
- Anterior Chamber Cell Count
- Anterior Chamber Cell Flare

#### Surgical Visit Day 0 First Eye

- Medical history and concurrent illnesses
- Concomitant medications
- Grade Cataract Density (scale 1 to 4)
- Indicate incision type, location, and size
- Type of IOL and lens power
- Record any surgical complications
- Subject reported AEs prior to or after surgery
- Insert intracanalicular dexamethasone insert (\*if randomized to Dextenza arm)
- Physician Ease of Use Survey
- Intracameral injection of NSAID+abx+steroid combo
- Insert visualization
- Prescribe post-operative regimen (\*specific to each eye)

## Day 1 First Eye (To be completed prior to 2<sup>nd</sup> eye sx)

- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- Slit lamp Exam
- IOP
- Subject reported AEs prior to or after surgery
- Ocular Pain Assessment

- Anterior Chamber Cell Count
- Anterior Chamber Cell Flare
- Insert visualization

#### Surgical Visit Day 0 Second Eye (To be completed one day after first eye sx)

- Medical history and concurrent illnesses
- Concomitant medications
- Grade Cataract Density (scale 1 to 4)
- Indicate incision type, location, and size
- Type of IOL and lens power
- Record any surgical complications
- Subject reported AEs prior to or after surgery
- Insert intracanalicular dexamethasone insert (\*if randomized to Dextenza arm)
- Physician Ease of Use Survey
- Intracameral injection of NSAID+abx+steroid combo
- Insert visualization
- Prescribe post-operative regimen (\*specific to each eye)

#### Day 1 Second Eye

- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- Slit lamp Exam
- IOP
- Subject reported AEs prior to or after surgery
- Ocular Pain Assessment
- Anterior Chamber Cell Count
- Anterior Chamber Cell Flare
- Insert visualization

#### Day 7 (+/- 2 days from first eye sx)

- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- MRX
- BCVA
- Slit lamp Exam
- IOP
- Subject reported AEs prior to or after surgery
- Eve Drop Burden Questionnaire
- Ocular Pain Assessment
- Anterior Chamber Cell Count

- Anterior Chamber Cell Flare
- Insert visualization

#### Day 28-35 (+/- 5 days from first eye sx)

- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- MRX
- BCVA
- Ophthalmic examination (dilated fundus exam)
- Slit lamp Exam
- OCT
- IOP
- Subject reported AEs prior to or after surgery
- Eye Drop Burden Questionnaire
- Adapted COMTOL Questionnaire
- Ocular Pain Assessment
- Anterior Chamber Cell Count
- Anterior Chamber Cell Flare
- Insert visualization

#### Month 3 (+/- 7 days from first eye sx)

- Medical history and concurrent illnesses
- Concomitant medications
- Distance VA
- BCVA
- Slit lamp Exam
- IOP
- Subject reported AEs prior to or after surgery
- Ocular Pain Assessment
- Anterior Chamber Cell Count
- Anterior Chamber Cell Flare
- Insert visualization

#### **Unscheduled Visits**

All attempts should be made to keep patients on the study schedule. Unscheduled visits may be necessary to repeat testing following abnormal laboratory results, for follow-up of AEs, or for any other reason, as warranted.

#### Adverse Event Information Collection

The investigator (or designee) will record all AEs that occur during the study The definition of an AE and SAE, and information on the determination of severity and relationship to treatment are provided in Section 6.

#### Rescue Criteria

- Patients should be rescued at any time at the discretion of the investigator.
- The following rescue criteria are to be applied by the investigator:
  - > Grade 3 anterior chamber cells
  - Ocular pain score of > 5 due to ocular inflammation
- Patients requiring rescue therapy will be prescribed: topical steroid and topical NSAID per the discretion of the investigator.

If a patient requires rescue therapy in the eye containing the dexamethasone insert, the insert will not be removed, and subjects will be followed for safety.

## Safety Definitions, Reporting, and Monitoring

#### **Definitions**

#### Adverse Event

An AE is any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug. Therefore, an AE is any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease which is temporally associated with the use of a study drug, whether or not considered related to the study drug.

An AE also includes any worsening (i.e. any clinically significant change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study drug.

#### Serious Adverse Event

A SAE is any untoward medical occurrence that at any dose:

- Results in **death** includes all deaths, even those that appear to be completely unrelated to study drug (e.g. a car accident in which a patient is a passenger).
- Is **life-threatening** in the view of the investigator, the patient is at immediate risk of death at the time of the event. This does not include an AE that had it occurred in a more severe form, might have caused death.
- Requires in-patient **hospitalization** or prolongation of existing hospitalization. In-patient hospitalization is defined as admission to a hospital or an emergency room for longer than 24 hours. Prolongation of existing hospitalization is defined as a hospital stay that is longer than

was originally anticipated for the event, or is prolonged due to the development of a new AE as determined by the investigator or treating physician.

- Results in persistent or significant **disability/incapacity** (substantial disruption of one's ability to conduct normal life functions).
- Is a congenital anomaly/birth defect
- Is an **important medical event** Important medical events may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the patient or may require intervention to prevent 1 of the other serious outcomes listed above (e.g., intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; or development of drug dependency or drug abuse). Any malignancy (other than basal cell skin cancers) would be considered a medically important event.

#### Recording and Reporting Adverse Events

All AEs and SAEs will be recorded only if they are medically relevant.

All SAEs, regardless of assessment of causal relationship to study insert will be reported to Ocular Therapeutix.

To report an SAE, Ocular Therapeutix will be contacted at the following:

ocutx.pharmacovigilance@propharmagroup.com

SAE hotline: 844-668-3948

The investigator will promptly report to the IRB all unanticipated problems involving risks to patients. This includes death from any cause and all SAEs related to the use of the study insert. All SAEs will be reported to the IRB, regardless of assessed causality.

## Study Variables

## Demographic and Baseline Characteristics

Baseline characteristics will include standard demography (e.g. age, race, weight, height, etc.), disease characteristics including medical history, and medication history for each patient.

## Ethical and Regulatory Considerations Good Clinical Practice Statement

It is the responsibility of the investigator(s) to ensure that this clinical study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki, and that are consistent with the ICH guidelines for Good Clinical Practice (GCP) and applicable regulatory requirements.

#### **Informed Consent**

The principles of informed consent are described in ICH Guidelines for GCP.

Ocular Therapeutix will have the right to review and comment on the informed consent form.

It is the responsibility of the investigator or designee (if acceptable by local regulations) to obtain written informed consent from each patient prior to his/her participation in the study and after the aims, methods, objectives, and potential hazards of the study have been explained to the patient in language that he/she can understand. The ICF will be signed and dated by the patient and by the investigator or authorized designee who reviewed the ICF with the patient.

Patients who can write but cannot read will have the ICF read to them before signing and dating the ICF.

Patients who can understand but who can neither write nor read will have the ICF read to them in presence of an impartial witness, who will sign and date the ICF to confirm that informed consent was given.

The original ICF will be retained by the investigator as part of the patient's study record, and a copy of the signed ICF will be given to the patient.

If new safety information results in significant changes in the risk/benefit assessment, the ICF will be reviewed and updated appropriately. All study patients will be informed of the new information and provide their written consent if they wish to continue in the study. The original signed revised ICF will be maintained in the patient's study record and a copy will be given to the patient.

## Patient Confidentiality and Data Protection

The investigator will take all appropriate measures to ensure that the anonymity of each study patient will be maintained.

The patient's and investigator's personal data will be treated in compliance with all applicable laws and regulations.

#### Institutional Review Board

An appropriately constituted IRB, as described in ICH Guidelines for GCP, will review and approve:

- The protocol, ICF, and any other materials to be provided to the patients (e.g. advertising) before any patient may be enrolled in the study
- Any amendment or modification to the study protocol or ICF before implementation, unless the change is necessary to eliminate an

immediate hazard to the patients, in which case the IRB will be informed as soon as possible

Ongoing studies will be reviewed by the IRB/EC on an annual basis or at intervals appropriate to the degree of risk.

In addition, the IRB will be informed of any event likely to affect the safety of patients or the continued conduct of the clinical study.

A copy of the IRB approval letter will be sent to Ocular Therapeutix prior to shipment of drug insert supplies to the investigator. The approval letter will include the study title, the documents reviewed, and the date of the review.

Records of the IRB review and approval of all study documents (including approval of ongoing studies) will be kept on file by the investigator.

#### **APPENDICES**

Protocol Appendix A: Ease of use Survey

Protocol Appendix B: Eye Drop Burden Questionnaire

Protocol Appendix C: Adapted COMTOL

#### REFERENCES

1. DEXTENZA [PACKAGE INSERT]. BEDFORD, MA: OCULAR THERAPEUTIX, INC; 2019.

- 2. Walters TR, Bafna S, Vold S, et al. Efficacy and Safety of Sustained Release Dexamethasone for the Treatment of Ocular Pain and Inflammation after Cataract Surgery: Results from Two Phase 3 Studies. *J Clin Exp Ophthalmol.* 2016;7(4):1-11.
- 3. Tyson SL, Bafna S, Gira JP, et al. Multicenter randomized phase 3 study of a sustained-release intracanalicular dexamethasone insert for treatment of ocular inflammation and pain after cataract surgery. [published correction appears in J Cataract Refract Surg. 2019;45(6):895]. J Cataract Refract Surg. 2019;45(2):204-212.

Protocol Appendix A: Ease of Use Survey

The investigator will grade the level of ease of insertion of the intracanalicular insert on a 0 to 10-point scale.

The Investigator will record ease of insertion procedure on the appropriate Case Report Form.

0 1 2 3 4 5 6 7 8 9 10

Very Easy

Very Hard

## Protocol Appendix B: **Eye Drop Burden Questionnaire**

| | | Never | Rarely | Sometimes | Usually | Always |
|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | 5 |
| 1. | I forget to administer my eye drops. | | | | | |
| 2. | It is difficult and/or frustrating to administer my eye drops. | | | | | |
| 3. | My eye drops<br>burn and/or sting<br>when I administer<br>them. | | | | | |
| 4. | My eye drop<br>treatment<br>interferes with the<br>daily activities of<br>my life. | | | | | |
| 5. | I forget to wash<br>my hands prior to<br>administering my<br>eye drops. | | | | | |
| 6. | I accidentally administer more and/or less than one eye drop to the eye. | | | | | |
| 7. | The drops miss<br>my eye when I<br>administer them. | | | | | |
| 8. | The bottle tip touches my eye when using my eye drops. | | | | | |
| | Add up the numbers Score. | for each sta | tement to ca | lculate the total | l Eye Drop B | Burden |
| | Total Eye Drop Bure | den Score = | | | | |
| | Low Eye Drop Burd<br>Moderate Eye Drop<br>High Eye Drop Burd | Burden: 19- | 29 | | | |

Protocol Appendix C: Adapted COMTOL

Comparison of Ophthalmic Medications for Tolerability (COMTOL) Questionnaire (adapted to compare physician & patient administered 'fewer-drops' regimen ((Treatment A- Experimental Group)) to patient-only administered total topical therapy ((Treatment B- Control Group)).

#### Interviewer: Please read the following verbatim!

Thank you for participating in our study. Your evaluation of the test "fewer-drops" treatment (Treatment A- Experimental Group) that the surgeon and you administered following your surgery compared to the total eyedrops (Treatment B- Control Group) you administered following surgery is most valuable to us. We would greatly appreciate your assistance by answering the following questions as best as possible. All answers are confidential.

Every patient received both treatment regimens. Every patient received Treatment A in one eye and Treatment B in the opposite eye. For clarification, here are the definitions of each treatment group:

#### Treatment A (Experimental Group-fewer-drops, physician & patient administered):

• Dextenza (steroid punctal plug/insert) + Vigamox drops 4x/day for 1st week + Prolensa drops 1x/day for one month

## **Treatment B (Control Group- total topical eyedrop therapy, patient-only administered):**

- Prednisolone drops 4x/day for 1<sup>st</sup> week, 3x/day for 2<sup>nd</sup> week, 2x/day for 3<sup>rd</sup> week, 1x/day for 4<sup>th</sup> week + Vigamox drops 4x/day for 1<sup>st</sup> week + Prolensa drops 1x/day for one month
- 1. (Interviewer: Questions 1 and 2 are to be asked only at the Month 1 Visit).

Now that you tried both test regimens, did you prefer the Treatment A (fewer-drops, physician & patient administered) regimen or the Treatment B (total eyedrop therapy, patient-only administered) regimen?

| (Interviewer: Please check the appropriate response below). | |
|-------------------------------------------------------------|----|
| Treatment A regimen (Experimental Group-fewer drops | 5) |
| Treatment B regimen (Control Group-all drops) | |
| Neither (Do not read) | |

2. Why did you prefer your selected treatment? (Interviewer: Read response from Question 1)

## 'Fewer-Drops' Physician/Patient-Administered Therapy (Treatment A): Patient Reported Outcomes

- 3. (Interviewer: Read the following). I am going to read to you a list of various side effects that may occur in some patients who receive Treatment A regimen ('fewer-drops' physician & patient administered regimen) following ophthalmic surgery. You may have experienced none, some, or all these side effects during the past month. As I read the list, please tell me if you experienced that side effect. (Interviewer: Check affirmative responses on the far left column of the list below Question #4. Place a check under the column marked "I did not have the symptom" below Question #4 for those symptoms not experienced by the patient. If patient experienced none of these side effects, please check "None of these symptoms" below and go to Question #6).
- 4. (Interviewer: Refer to Question #3 and read the following). I am now going to read to you the side-effects you said you experienced in the last question. For each side effect I mention, please tell me how frequently you experienced each side effect during the past month. (interviewer- hand respondent Card "A" with frequency scales.) That is, did you experience the side effect rarely, a few times, often, use ally, almost always, or always? (Interviewer: Place check under appropriate column below for each checked side effect mentioned by respondent).

| | | Hav | Not<br>e the<br>ptom | Rar | <u>ely</u> | | A Few<br>Times | | <u>Fairly</u><br><u>Often</u> | | <u>Usually</u> | | Almost<br>Always | | vays_ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Burning/stinging in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Redness in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Blurred vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Bitter taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Unusual taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Itchy eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Discharge from eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Swelling of eyelids | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Brow ache | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dimming of vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Difficulty in focusing from near to far | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dry eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Trouble reading | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Trouble seeing at night | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Tearing | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | None of these symptoms | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |

5. (Interviewer: Refer to Question #4 and read the following). I am again going to repeat the side-effects you just mentioned. For each side effect I mention, please tell me if you have been bothered by it: not at all, a little, some, quite a bit, very much so, or extremely so? (Interviewer: Place check under appropriate columns below)

| | | Not | at all | <u>A 1</u> | <u>ittle</u> | So | Some | | Quite a bit | | Very much so | | nely so |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Burning/stinging in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Redness in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Blurred vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Bitter taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Unusual taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Itchy eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Discharge from eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Swelling of eyelids | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Brow ache | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dimming of vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Difficulty in focusing from near to far | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dry eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Trouble reading | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Trouble seeing at night | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Tearing | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |

6. During the past month has your quality of life been interfered with by these side effects: not at all, a little, some, quite a bit, very much so, or extremely so?

| <br>N | ot | at | all |
|-------|-----|----|-----|
| | 4 . | 4 | |

A little Some

Quite a bit

Very much so

Extremely so

7. (Interviewer). I am now going to show you a list of activities you might do during a typical day. You may perform none, some, or all of these activities. For each one on the list, please tell me whether you perform it on a routine basis. (Interviewer: Hand

| | hose | | | | | | • | elow th<br>Card | | menti | oned by |
|---|---|---|---|---|---|---|---|---|---|---|---|
| eries | | | | | | | | | | | |
| rs | | | | | | | | | | | |
| lewspa | per | | | | | | | | | | |
| one, ponth le physery much | lease<br>becau<br>sician<br>ch so, | tell ruse of | ne if<br>the<br><b>atie</b> i | you<br>Treant). I | were<br>t <b>me</b><br>That | e limitent A | ted at<br>r <b>egin</b><br>re yo | all in<br>en (fe<br>u limit | perform<br>wer-d<br>ted: no | ming e rops r ot at al | ach<br><b>egimen</b><br>l, a little |
| Not | at all | <u>A 1</u> | <u>ittle</u> | Sc | <u>me</u> | Quite | a bit | Very n | nuch so | Extre | nely so |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ; ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| in perf | | _ | • | | | | | | | _ | n<br>nth, has |
| | now gone, pononth le physery much below | newspaper now going one, please month because physician ery much so, a below) Not at all ( ) ( ) ( ) ( ) ( ) ( ) | newspaper now going to recone, please tell recone, please tell recone are physician & pery much so, or enter below) Not at all All () (() () | newspaper now going to repeat one, please tell me if month because of the rephysician & patient a below) Not at all A little ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) | newspaper now going to repeat each one, please tell me if you month because of the Treate physician & patient). The ery much so, or extremely to below) Not at all A little Some () | newspaper I now going to repeat each of tone, please tell me if you were month because of the <b>Treatmente physician &amp; patient</b> ). That ery much so, or extremely so? In below) Not at all A little Some ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) | newspaper I now going to repeat each of the act one, please tell me if you were limit month because of the <b>Treatment A</b> is the physician & patient). That is, we try much so, or extremely so? (Internabelow) Not at all A little Some Quite () | newspaper I now going to repeat each of the activities one, please tell me if you were limited at month because of the <b>Treatment A regin te physician &amp; patient</b> ). That is, were your much so, or extremely so? (Interview on below) Not at all A little Some Quite a bit ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) ( ) | newspaper I now going to repeat each of the activities you jone, please tell me if you were limited at all inmonth because of the Treatment A regimen (few physician & patient). That is, were you limitery much so, or extremely so? (Interviewer: Please below) Not at all A little Some Quite a bit Very many (a) (a) (b) (b) (c) (c | newspaper I now going to repeat each of the activities you just sail one, please tell me if you were limited at all in performanth because of the Treatment A regimen (fewer-die physician & patient). That is, were you limited: not retry much so, or extremely so? (Interviewer: Please charbelow) Not at all A little Some Quite a bit Very much so () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () () | newspaper In now going to repeat each of the activities you just said you one, please tell me if you were limited at all in performing emonth because of the Treatment A regimen (fewer-drops rephysician & patient). That is, were you limited: not at all ery much so, or extremely so? (Interviewer: Please check of just below) Not at all A little Some Quite a bit Very much so Extremely in the little of the l |

#### Total Topical Eyedrop therapy patient-administered: Patient Reported Outcomes

- 10. (Interviewer: Read the following). I am going to read to you a list of various side effects that may occur in some patients who receive Treatment B (self-administered total eyedrop therapy following ophthalmic surgery). You may have experienced none, some, or all these side effects during the past month. As I read the list, please tell me if you experienced that side effect. (Interviewer: Circle affirmative responses on the list below. Place a check under the column marked "I did not have the symptom" below for those symptoms not experienced by the patient. If patient experienced none of these side effects, please check "None of these symptoms" below and go to Question # 10).
- 11. (Interviewer: Refer to Question #7 and read the following). I am now going to read to you the side-effects you said you experienced in the last question. For each side effect I mention, please tell me how frequently you experienced each side effect during the past month. (interviewer- hand respondent Card "A" with frequency scales.) That is, did you experience the side effect rarely, a few times, often, usually, almost always, or always? (Interviewer: Place check under appropriate column below for each circled side effect mentioned by respondent).

| | | | d Not<br>e the<br>ptom | Rai | rel <u>y</u> | | rew<br>nes | | <u>Fairly</u><br><u>Often</u> | | <u>Usually</u> | | Almost<br>Always | | <u>vays</u> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Burning/stinging in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Redness in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Blurred vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Bitter taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Unusual taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Itchy eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Discharge from eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Swelling of eyelids | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Brow ache | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dimming of vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Difficulty in focusing from near to far | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dry eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Trouble reading | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Trouble seeing at night | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Tearing | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | None of these symptoms | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |

| <i>12</i> . | (Interviewer: Refer to Question #7 and read the following). I am again going to repeat |
|---|---|
| | the side-effects you just mentioned. For each side effect I mention, please tell me if you have |
| | been bothered by it: not at all, a little, some, quite a bit, very much so, or extremely so? |
| | (Interviewer: Place check under appropriate columns below) |

| | | Not | at all | <u>A 1</u> | <u>ittle</u> | So | Some | | a bit | Very n | nuch so | Extremely so | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Burning/stinging in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Redness in eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Blurred vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Bitter taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Unusual taste | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Itchy eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Discharge from eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Swelling of eyelids | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Brow ache | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Dimming of vision | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Difficulty in focusing from near to far | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Dry eyes | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Trouble reading | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| _ | Trouble seeing at night | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |
| | Tearing | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) | ( | ) |

13. During the past month has your quality of life been interfered with by these side effects: not at all, a little, some, quite a bit, very much so, or extremely so?

| Not at all |
|------------------|
| A little |
| Some |
| Quite a bit |
| Very much so |
| <br>Extremely so |

| Dri<br>Lif<br>Cli<br>Wa<br>Rea | iving during the day iving at night fing or carrying grocers alking 1 flight of stairs alking several blocks ading the newspaper ading other than the newspaper activity in the past more iving the past more interest. | wspa<br>now g<br>ne, pl | oing | tell r | ne if | you | were | e limi | ed at | all in | perfor | ming e | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | | | my much |
| | administered). That is so, or extremely so? ( | Inter | viewe | er: P | lease | che | ck oj | ff und | ler ap | propr | iate co | lumn | below) |
| | administered). That is so, or extremely so? ( | Inter | - | er: P | | che | ck oj | ff und | ler ap | propr | - | lumn | • |
| _ | administered). That | Inter | viewe<br>at all | er: P | lease<br>ittle<br>) | So ( | c <b>k o</b> j<br>me<br>) | ff und<br>Quite | ler ap<br>a bit | Very n | iate co | lumn | below) |
| | administered). That is so, or extremely so? ( Driving during day Driving at night Lifting or carrying | Inter | viewe | er: P | lease | So ( | ck oj | ff und<br>Quite | ler ap | Very n | iate co | lumn | below) |
| | administered). That is so, or extremely so? ( | Inter | viewe<br>at all | er: P | lease<br>ittle<br>) | So ( | c <b>k o</b> j<br>me<br>) | ff und<br>Quite | ler ap<br>a bit | Very n | iate co | lumn | below) |
| | administered). That is so, or extremely so? ( Driving during day Driving at night Lifting or carrying groceries | Inter | viewe<br>at all | er: P | lease<br>ittle<br>) | So ( | c <b>k o</b> j<br>me<br>) | ff und<br>Quite | ler ap<br>a bit | Very n | iate co | lumn | below) |
| | administered). That is so, or extremely so? ( Driving during day Driving at night Lifting or carrying groceries Climbing 1 flight of stairs | Inter | viewe<br>at all | er: P | lease<br>ittle<br>) | So ( | c <b>k o</b> j<br>me<br>) | ff und<br>Quite | ler ap<br>a bit | Very n | iate co | lumn | below) |

| The PREPARE Study (V1) |
|---|
| A little Some Quite a bit Very much so Extremely so |
| 17. During the past month, how often did you miss one or more doses of the eyedrop medication? |
| I did not miss any doses |
| Rarely |
| A few times Fairly often |
| Usually |
| Almost always |
| Always |
| <ul> <li>18. Overall, how satisfied, if at all, have you been with the regimen you stated you preferred? (Interviewer: Hand respondent Card C with satisfaction scales) Would you say you were totally satisfied, very satisfied, somewhat satisfied, somewhat dissatisfied, very dissatisfied or totally dissatisfied? (Interviewer: Record only one response below)</li> <li>Totally satisfied</li> <li>Very satisfied</li> <li>Somewhat satisfied</li> <li>Somewhat dissatisfied</li> <li>Very dissatisfied</li> <li>Totally dissatisfied</li> </ul> |
| Thank respondent and terminate interview. |
| Signature of Interviewer Date |

Very satisfied

Somewhat satisfied

Very dissatisfied

Totally dissatisfied

Somewhat dissatisfied

## Card A I did not have the symptom Rarely A few times Fairly often Usually Almost always Always Card B Driving during the day Driving at night Lifting or carrying groceries Climbing 1 flight of stairs Walking several blocks Reading the newspaper Reading other than the newspaper Card C Totally satisfied